CLINICAL TRIAL: NCT06128330
Title: Point-of-care Measurement of the Antifibrinolytic Activity of Tranexamic Acid in Cardiac Surgery
Acronym: PAATICS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-02070
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Antifibrinolytic Agents
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dose group (Active Comparator): The standard dose group will receive a bolus of 20 mg/kg tranexamic acid after anaesthesia induction.
  Interventions: Drug: Tranexamic acid bolus 20 mg/kg
- Low dose group (Experimental): The low dose group will receive a bolus of 10 mg/kg tranexamic acid. In addition 1 mg/kg tranexamic acid will be added to the priming of the extracorporeal circuit (ECC) and a continuous infusion of 1mg/kg/h tranexamic acid will be started after the bolus infusion until the end of surgery.
  Interventions: Drug: Tranexamic acid bolus 10 mg/kg; Drug: Tranexamic acid bolus 1 mg/kg; Drug: Tranexamic acid continuous infusion of 1 mg/kg/h in the low dose group

INTERVENTIONS:
Drug: Tranexamic acid bolus 20 mg/kg — Bolus of tranexamic acid in the standard dose group
  Arms: Standard dose group
Drug: Tranexamic acid bolus 10 mg/kg — Bolus of tranexamic acid in the low dose group
  Arms: Low dose group
Drug: Tranexamic acid bolus 1 mg/kg — Bolus of tranexamic acid in the low dose group (to add into the CPB prime)
  Arms: Low dose group
Drug: Tranexamic acid continuous infusion of 1 mg/kg/h in the low dose group — Tranexamic acid continuous infusion during the procedure
  Arms: Low dose group

SUMMARY:
Tranexamic acid (TXA) is a widely used antifibrinolytic agent that can reduce postoperative blood loss and packed red blood cell transfusions during cardiac surgery. Previous (in-vivo) studies have measured TXA plasma concentration and associated clinical effect (e.g. blood loss). Patient blood management guidelines recommend the routine use of TXA in cardiac surgery, especially for procedures with a high risk of bleeding.

A new point-of-care viscoelastic diagnostic assay (tissue plasminogen activator assay, TPA assay) allows for a rapid determination of antifibrinolytic activity in a patient in the operating room making TXA dose adjustment easily possible intraoperatively. Currently, there is no consensus on the dosing of TXA and different protocols are used. Recommendations for high doses (e.g. 30 mg/kg followed by 16 mg/kg per hour during cardiac surgery with 2 mg/kg added to extracorporeal circulation) alternate with recommendations for low doses (e.g., 10 mg/kg followed by 1 mg/kg per hour for 12 hours).

Tranexamic acid administration increases the risk of postoperative seizure, a risk that appears to be dose dependant. A recent meta-analysis suggests that a single TXA bolus of 20 mg/kg is sufficient to reduce postoperative blood loss and packed red blood cell transfusion in patients undergoing aortocoronary bypass surgery. The calculations in the meta-analysis were, however, based on a simulation of blood concentrations of TXA by a pharmacokinetic model, so the results are subject to many uncertainties. The optimal TXA regimen for cardiac surgery, both in terms of efficacy and safety therefore remains uncertain and requires further investigation.

This study was invented to determine the actual levels of tranexamic acid in vivo to observe antifibrinolytic activity during cardiac surgery up to 48 hours after termination of surgery. The risk category is evaluated as risk category A as the study is a clinical trial examining the effect of drugs that are already authorized for the clinical use.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients:

* Over 18 years old
* Elective surgery
* Written informed consent
* Patient planned for aortocoronary artery bypass graft surgery, aortic valve replacement or mitral valve surgery (or a combination of these procedures)
* Normal renal function
* No previous intake of anticoagulants except acetylsalicylic acid in the preoperative period

Exclusion Criteria:

* Impaired renal function (eGFR < 30 ml/min.)
* History of seizure
* Pregnancy
* Inability to understand and sign the informed consent (e.g., language problems, dementia, psychological disorders)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
TPA test | 48 hours after completion of surgery
  The primary endpoint of the study is if the antifibrinolytic activity as measured with the TPA assay. The result can be positive (no fibrinolysis and good antifibrinolytic activity) or negative (fibrinolysis and no antifibrinolytic activity).The TPA assay is performed at five different time points until the 2. postoperative day (48 hours).

SECONDARY OUTCOMES:
Chromatography | 48 hours after completion of surgery
  Secondary endpoint is the TXA concentration as measured by chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kauert-Willms, MD, Principal Investigator — University Hospital Berne
Locations (1):
- Dpt. Anesthesiology and pain Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No